CLINICAL TRIAL: NCT07022210
Title: Incidence of Hypotension in the Post-anesthesia Care Unit (PACU).
Status: Recruiting | Type: Observational
Sponsor: Tomas Bata Hospital, Czech Republic (Other)
Responsible Party: Principal Investigator, Klára Nekvindová, Deputy Chief for Science, Education, and Research, Tomas Bata Hospital, Czech Republic
Other Study IDs: 2025-12
Record Dates: First submitted 2025-05-22; First posted 2025-06-15 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Hypotension During Surgery; Surgery-Complications
Keywords: hypotension; post-anesthesia care unit; surgery; adult
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The perioperative period poses a heightened risk of complications for patients, including hypotension. While the issue of intraoperative hypotension is well-documented in medical literature, the occurrence and causes of hypotension in the post-anesthesia care unit often receive less attention. This phase of postoperative care, however, is vital for ensuring patient stability and preventing severe consequences. Failure to identify and manage a drop in blood pressure can lead to hypoperfusion of critical organs, increasing the risk of morbidity and mortality. The aim of this study is to examine the frequency of hypotension in the post-anesthesia care unit-defined as systolic blood pressure <90 mmHg or a drop of more than 20% from baseline-and to identify factors contributing to its development.

DETAILED DESCRIPTION:
The perioperative period is a critical time for patients, marked by an increased risk of various complications, including hypotension. While intraoperative hypotension is extensively studied in medical literature, the occurrence and underlying causes of hypotension in the post-anesthesia care unit (PACU) often remain overlooked. This phase of postoperative care is essential for stabilizing the patient and preventing severe outcomes. A failure to identify and adequately address a drop in blood pressure during this time can result in hypoperfusion of vital organs, increasing the likelihood of morbidity and mortality.

Hypotension in the PACU is defined as a systolic blood pressure below 90 mmHg or a decrease exceeding 20% compared to the patient's baseline measurements. The aim of this research is to explore the prevalence of hypotension in the PACU and to analyze the factors contributing to its occurrence. By improving the understanding of this issue, the study seeks to enhance patient outcomes through timely identification and management of hypotension in this crucial phase of care.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* patients undergoing a procedure under general anesthesia
* patients who have consented to data processing
* postoperative stay in PACU

Exclusion Criteria:

* patients younger than 18 years old.
* patients transferred directly to the ICU/Anesthesiology and Resuscitation Department after surgery without staying in the recovery room.
* patients with incomplete medical documentation or missing blood pressure values in the recovery room.
* patients with a pre-existing diagnosis of resistant hypotension or unstable hemodynamics before surgery
* patients with a history of long-term use of anxiolytics, antipsychotics, or other psychotropic medications that may affect cognitive function, emotional state, or predictive outcomes
* patient refusal to participate in the study (including cases where they initially consented), with an emphasis on respecting patient autonomy

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients meeting the inclusion criteria, aged 18 to 105 years, with an indicated hospitalization at a diagnostic-therapeutic unit (DTU).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypotension in the post-anesthesia care unit (PACU). | 0. postoperative day
  Hypotension is defined as systolic blood pressure <90 mmHg or a decrease of more than 20% from baseline values.

SECONDARY OUTCOMES:
Duration of the operation | 0. postoperative day
  Duration of the surgical procedure as a risk factor for the development of postoperative hypotension. The duration will be recorded in minutes.
ASA classification (American Society of Anesthesiologists classification). | 0. postoperative day
  ASA classification as a risk factor for the development of postoperative hypotension.
  ASA I: A normal healthy patient with no systemic disease. ASA II: A patient with mild systemic disease that does not limit daily activities (e.g., well-controlled diabetes or hypertension).
  ASA III: A patient with severe systemic disease that limits daily activities but is not incapacitating (e.g., poorly controlled diabetes or hypertension, chronic obstructive pulmonary disease).
  ASA IV: A patient with severe systemic disease that is a constant threat to life (e.g., unstable angina, symptomatic heart failure).
  ASA V: A moribund patient who is not expected to survive without surgery (e.g., ruptured abdominal aneurysm).
Type of anesthesia. | 0. postoperative day
  The type of anesthesia used: general, regional, and/or peripheral nerve block.
Blood loss during the operation | 0. postoperative day
  Blood loss during the surgical procedure, as documented in the surgical protocol.
Fluid balance during the surgery | 0. postoperative day
  Fluid intake and output during surgery, measured in milliliters.
Surgical specialty | 0. postoperative day
  Surgical specialties: neurosurgery, urology, gynecology, abdominal surgery, orthopedics
Fluid administration in the recovery room. | 0. postoperative day
  Administration of a crystalloid or colloid bolus to augment intravascular volume.
Administration of vasopressors. | 0. postoperative day
  In cases of severe hypotension, vasopressor administration (e.g., ephedrine, phenylephrine, norepinephrine) may be required to ensure adequate perfusion of vital organs.
Blood pressure monitoring. | 0. postoperative day
  Repeated blood pressure measurement every 5 minutes.
Heart rate monitoring. | 0. postoperative day
  Continuous heart rate monitoring.
Patient repositioning | 0. postoperative day
  The Trendelenburg position (legs elevated above the head) can help increase venous return and consequently blood pressure. It will not be performed in surgeries involving the lower extremities.
Transfer of the patient to the ICU due to hemodynamic instability | 0. postoperative day
  If hypotension does not improve despite repeated therapeutic interventions, escalation of care to the ICU may be necessary.
Postoperative nausea and vomiting | 0. postoperative day
  Inadequate gastrointestinal perfusion can lead to nausea and vomiting, complicating the patient's recovery.
Impaired diuresis (oliguria, anuria) | 0. postoperative day
  Oliguria is a medical term referring to low urine output, typically defined as producing less than 400-500 mL of urine per day in adults.
  Anuria is a medical condition characterized by the absence or near absence of urine production, typically defined as less than 100 mL of urine per day.
Impaired consciousness - GCS | 0. postoperative day
  The Glasgow Coma Scale (GCS) is a clinical tool used to assess a person's level of consciousness after a brain injury. It evaluates three responses: eye opening, verbal response, and motor response, with scores ranging from 3 (deep coma) to 15 (fully alert).
Hypoxia | 0. postoperative day
  Will be assessed using oxygen saturation levels (SpO₂). Mild hypoxia: SpO₂ 90-94% Moderate hypoxia:r SpO₂ 75-89% Severe hypoxia: SpO₂ <75%
Lactic acidosis | 0. postoperative day
  Lactic acidosis is a condition characterized by the accumulation of lactic acid in the bloodstream, leading to a decrease in blood pH. It can result from tissue hypoxia, impaired metabolism, or certain medical conditions.
  Lactic acidosis is generally defined by a serum lactate concentration above 4 mmol/L. Mild elevations in lactate (hyperlactatemia) occur at levels above 2 mmol/L, but true lactic acidosis is diagnosed when lactate levels exceed 4 mmol/L
Syncope | 0. postoperative day
  Syncope is a temporary loss of consciousness due to a sudden decrease in blood flow to the brain. It typically has a rapid onset, short duration, and spontaneous recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Tomas Bata regional Hospital, Zlín, Czechia

IPD SHARING:
Plan to Share IPD: Undecided